CLINICAL TRIAL: NCT00889681
Title: CAP-AF: Continued Access Protocol for the Evaluation of Catheter Cryoablation in the Treatment of Paroxysmal Atrial Fibrillation
Brief Title: Continued Access Protocol
Acronym: CAP-AF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAP PS-024
Record Dates: First submitted 2009-04-24; First posted 2009-04-29 (Estimated); Results first posted 2014-04-25 (Estimated); Last update posted 2018-09-19 (Actual); Status verified 2018-09

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ablation (Experimental): All study subjects will be receive cryo ablation with the experimental devices and, optionally, an Atrial Fibrillation Drug.
  Interventions: Device: Arctic Front Cardiac Cryoablation System

INTERVENTIONS:
Device: Arctic Front Cardiac Cryoablation System — The CryoCath Arctic Front® Cardiac CryoAblation Catheter System, including the Freezor MAX Cardiac Cryoablation Catheter, is indicated for the treatment of patients with paroxysmal atrial fibrillation to reduce the likelihood of subsequent detectable atrial fibrillation.
  Other Names: Arctic Front® Catheter Ref# 2AF232 & 2AF282; Manual Retraction Kit Ref# 20MRK; Freezor MAX Catheter Ref # 239F3 & 239F5; Console Ref # 106A2

SUMMARY:
This Continued Access Protocol has been written to allow ongoing treatment of subjects at selected investigational sites while the marketing application for the Arctic Front® Cryoablation System is under review. This study will also allow collection of additional safety data following modifications implemented into the Arctic Front® Catheter and Cryoablation System.

DETAILED DESCRIPTION:
1. To evaluate the safety of treatment with the Arctic Front® Cardiac CryoAblation Catheter System, including the Freezor® MAX Cardiac Cryoablation Catheter by assessing the continuous survival of subjects free from one or more primary safety outcome measures-Cryoablation Procedure Events (CPEs) and Major Atrial Fibrillation Events (MAFEs), in adult patients with paroxysmal atrial fibrillation who have failed one or more Atrial Fibrillation Drugs (AFDs).
2. To evaluate the effectiveness of treatment with the Arctic Front® Cardiac CryoAblation Catheter System, including the Freezor® MAX Cardiac Cryoablation Catheter by assessing the continuous survival of subjects with success in the primary effectiveness outcome measure of Long Term Clinical Success (LTCS) in adult patients with paroxysmal atrial fibrillation who have failed one or more Atrial Fibrillation Drugs (AFDs).
3. To evaluate the acute performance of the modified Arctic Front® Cardiac CryoAblation Catheter System for comparison with the Arctic Front® Cardiac CryoAblation Catheter System used in the PS-023 STOP AF Pivotal Trial.

ELIGIBILITY:
Inclusion Criteria:

Subjects must fulfill ALL of the following criteria:

1. Documented PAF:

   * diagnosis of paroxysmal atrial fibrillation (PAF) (Section 9.1.18, General Protocol Terminology), AND
   * 2 or more episodes of AF during the 3 months preceding the Consent Date, at least 1 of which must be documented with a tracing
2. 18 and 75 years of age
3. Failure for the treatment of AF (effectiveness or intolerance) of one or more of the following drugs indicated in the treatment of PAF: flecainide, propafenone, sotalol or dofetilide.

Exclusion Criteria:

ANY of the following is regarded as a criterion for excluding a subject from the study:

1. Any previous left atrial (LA) ablation (except permissible retreatment subjects)
2. Any previous LA surgery
3. Current intracardiac thrombus (can be treated after thrombus is resolved)
4. Presence of any pulmonary vein stents
5. Presence of any pre-existing pulmonary vein stenosis
6. Pre-existing hemidiaphragmatic paralysis
7. Anteroposterior LA diameter > 5.5 cm by TTE
8. Presence of any cardiac valve prosthesis
9. Clinically significant mitral valve regurgitation or stenosis
10. Myocardial infarction, PCI / PTCA or coronary artery stenting which occurred during the 3 month interval preceding the Consent Date
11. Unstable angina
12. Any cardiac surgery which occurred during the 3 month interval preceding the Consent Date
13. Any significant congenital heart defect corrected or not (including atrial septal defects or pulmonary vein abnormalities but not including minor PFO)
14. NYHA class III or IV congestive heart failure
15. Left ventricular ejection fraction (LVEF) < 40%
16. 2º (Type II) or 3º atrioventricular block
17. Presence of a permanent pacemaker, biventricular pacemaker, atrial defibrillator or any type of implantable cardiac defibrillator (with or without biventricular pacing function)
18. Brugada syndrome
19. Long QT syndrome
20. Arrhythmogenic right ventricular dysplasia
21. Sarcoidosis
22. Hypertrophic cardiomyopathy
23. Known cryoglobulinemia
24. Uncontrolled hyperthyroidism
25. Any cerebral ischemic event (strokes or TIAs) which occurred during the 6 month interval preceding the Consent Date.
26. Any woman known to be pregnant
27. Any woman without freedom from pregnancy as demonstrated by one or more of the following conditions:

    * negative β-HCG test within 7 days prior to Start Date
    * history of surgical sterilization
    * postmenopausal and free of menses for at least 12 months.
28. Life expectancy less than one (1) year
29. Current or anticipated participation in any other clinical trial of a drug, device or biologic during the duration of this study
30. Unwilling or unable to comply fully with study procedures and follow-up

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2009-03; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Packer, MD, Principal Investigator — Mayo Clinic, Rochester, MN
Locations (10):
- United States (10):
  - Banner Good Samaritan, Phoenix, Arizona
  - Cedars Sinai Medical Center, Los Angeles, California
  - Stanford Hospital & Clinical, Stanford, California
  - Bay Heart Group, Tampa, Florida
  - Piedmont Hospital, Atlanta, Georgia
  - Massachusetts General Hospital, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Baylor Heart & Vascular Hospital, Dallas, Texas
  - Inova Research Center, Falls Church, Virginia
  - Virginia Commonwealth University Health System, Richmond, Virginia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Investigators at ten (10) sites enrolled a total of 81 study subjects between March 31, 2009 and January 24, 2011. The first subject was cryoablated on April 3, 2009.
Pre-assignment Details: There were three (3) subjects who were early exits in the study, two for not meeting qualification criteria and one for insurance disapproval.
Groups:
- Enrolled for Cryoablation Treatment: All patients that signed the informed consent were considered enrolled. Patients enrolled in the study received cryoablation treatment for paroxysmal atrial fibrillation.
Period: Overall Study
Arm/Group | Enrolled for Cryoablation Treatment
Started | 81
Received Treatment | 78
Completed | 78
Not Completed | 3
Not completed — Not meeting qualification Criteria | 2
Not completed — Insurance disapproval | 1

BASELINE CHARACTERISTICS:
Population: All enrolled subjects
Groups:
- Enrolled for Cryoablation Treatment: All patients that signed the informed consent were considered enrolled. Patients enrolled in the study to receive cryoablation treatment for paroxysmal atrial fibrillation.
Arm/Group | Enrolled for Cryoablation Treatment
Number analyzed (Participants) | 81
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 56
  >=65 years | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.7 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 59
Region of Enrollment [Number; unit: participants]
  United States | 81

OUTCOME MEASURES:

1. Primary Outcome: Cryoablation Procedure Events (CPEs)
Description: Composite event: access site complications, cardiac damage (including myocardial infarction), embolic phenomena (including stroke), arrhythmia, persistent phrenic nerve injury, death and pulmonary vein stenosis.
Time Frame: 365 days
Population: 78 of the 81 enrolled subjects were treated with cryoablation.
Measure: Number; unit: Participants
Groups:
- Treated With Cryoablation: Enrolled patients that underwent a cryoablation procedure for the treatment of paroxysmal atrial fibrillation.
Arm/Group | Treated With Cryoablation
Number analyzed (Participants) | 78
Participants
  One or more CPE (all types) | 1
  CPE type: Access site complications | 0
  CPE type: Cardiac damage (including MI) | 0
  CPE type: Embolic phenomena (including stroke) | 0
  CPE type: Arrhythmias | 1
  CPE type: Persistent phrenic nerve injury | 0
  CPE type: Death | 0
  CPE type: Pulmonary vein stenosis | 0

2. Primary Outcome: Acute Procedural Success (APS)
Description: Demonstration of electrical isolation in ≥ 3 pulmonary veins or their anomalous equivalents at the conclusion of the first protocol-defined cryoablation procedure.
Time Frame: At the conclusion of the cryoablation procedure
Population: 78 of 81 subjects were treated with cryoablation.
Measure: Number; unit: Participants
Arm/Group | Treated With Cryoablation
Number analyzed (Participants) | 78
Participants | 75

3. Primary Outcome: Freedom From Major Atrial Fibrillation Events (MAFE)
Description: Composite event including: cardiovascular death, hospitalization for: (AF recurrence or ablation, atrial flutter ablation (excluding Type I), systemic embolization (not stroke), congestive heart failure, hemorrhagic event (not stroke)), anti-arrhythmic drug: initiation, adjustment or complication, myocardial infarction, stroke.
Time Frame: 365 days
Population: 78 of 81 enrolled subjects were treated with cryoablation.
Measure: Number; unit: Participants
Arm/Group | Treated With Cryoablation
Number analyzed (Participants) | 78
Participants
  Freedom from any MAFE (all types) | 74
  One or more MAFE (all types) | 4
  MAFE type: Cardvascular death | 0
  MAFE type: Hosp for AF recurrence or ablation | 2
  MAFE type: Hosp for A flutter ablation (ex Type I) | 0
  MAFE type: Hosp for systemic embolism (not stroke) | 0
  MAFE type: Hosp for congestive heart failure | 0
  MAFE type: Hosp for hemorrhagic event (not stroke) | 2
  MAFE type: Antiarrhythmic medication | 1
  MAFE type: Myocardial infarction | 0
  MAFE type: Stroke | 0

4. Primary Outcome: Long-term Clinical Success
Description: Composite of both Acute Procedural Success and freedom from Chronic Treatment Failure. Freedom from Chronic Treatment Failure (CTF) was defined as no occurrence of an AF Intervention and no occurrence of Detectable AF which is defined as an episode of AF, documented in a tracing, and lasting more than 30 seconds, occurring during a Non Blanked Follow-up Period.
Time Frame: 180 days
Population: 78 of 81 subjects were treated with cryoablation.
Measure: Number; unit: Participants
Arm/Group | Treated With Cryoablation
Number analyzed (Participants) | 78
Participants | 51

ADVERSE EVENTS:
Time Frame: From time of consent to study exit (mean follow up time 3.4 years)
Description: Serious Adverse Event: a) resulting in death, b) life-threatening, c) resulting in inpatient hospitalization >48 hrs or prolongation of existing hospitalization by 2 or more days, d) resulting in persistent, significant, disability or incapacity, or e) resulting in a congenital anomaly or birth defect.
Groups:
- Treated With Cryoablation: This study is a single arm, non-randomized controlled study of patients with PAF referred for ablation after failing one or more antiarrhythmic drugs used in the treatment of AF ("Atrial Fibrillation Drugs " or AFDs). All study subjects will be receiving cryoablation with the experimental devices and, optionally, an Atrial Fibrillation Drug.
  Arctic Front Cardiac Cryoablation System : The CryoCath Arctic Front® Cardiac CryoAblation Catheter System, including the Freezor MAX Cardiac Cryoablation Catheter, is indicated for the treatment of patients with paroxysmal atrial fibrillation to reduce the likelihood of subsequent detectable atrial fibrillation.
Arm/Group | Treated With Cryoablation
Serious Adverse Events (participants affected / at risk) | 12/78
Other Adverse Events (participants affected / at risk) | 33/78
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treated With Cryoablation (N=78)
Atrial Fibrillation (Cardiac disorders) | 6 (8)
Drug Therapy (Surgical and medical procedures) | 1 (2)
Atrial Flutter (Cardiac disorders) | 1 (1)
Bladder Repair (Surgical and medical procedures) | 1 (1)
Bleeding Duodenal Ulcer (Gastrointestinal disorders) | 1 (1)
Cardiac Tamponade (Cardiac disorders) | 1 (1)
Cerebrovascular Accident (Nervous system disorders) | 1 (1)
Dizziness (Cardiac disorders) | 1 (1)
INR ratio increased (Blood and lymphatic system disorders) | 1 (1)
Migraine (Vascular disorders) | 1 (1)
Orchitis (Reproductive system and breast disorders) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Acute Renal Failure (Renal and urinary disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treated With Cryoablation (N=78)
CATHETER SITE HAEMATOMA (General disorders) | 11 (16)
PALPITATIONS (Cardiac disorders) | 8 (11)
ATRIAL FLUTTER (Cardiac disorders) | 7 (9)
ATRIAL FIBRILLATION (Cardiac disorders) | 7 (9)
CATHETER SITE HAEMORRHAGE (General disorders) | 7 (9)
NAUSEA (Gastrointestinal disorders) | 7 (7)
COUGH (Respiratory, thoracic and mediastinal disorders) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No